CLINICAL TRIAL: NCT06388343
Title: Causes of Listening Difficulties in Children
Acronym: CLINIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: S68485
Record Dates: First submitted 2024-04-18; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Listening Difficulties
Keywords: Listening difficulties; Multidisciplinary behavioral assessment; ECLiPS; Profiles

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with listening difficulties (Experimental): Comorbid developmental disorders Longitudinal study design (3 years) ECLiPS-questionnaire + behavioral measures
  Interventions: Other: Evaluation of Children's Listening and Processing Skills; Behavioral: Multidisciplinary behavioral assessment
- Typically developing children (Active Comparator): TD children perform the same behavioral tasks and ECLiPS-questionnaire to determine cut-off criteria for establishing a diagnosis.
  Interventions: Other: Evaluation of Children's Listening and Processing Skills; Behavioral: Multidisciplinary behavioral assessment

INTERVENTIONS:
Other: Evaluation of Children's Listening and Processing Skills — The Evaluation of Children's Listening & Processing Skills (ECLiPS; (Barry & Moore, 2021; Barry et al., 2015; Petley et al., 2021) is a caregiver-report outcome measure to profile auditory and cognitive real-world abilities important for successful listening and (auditory) processing.
  Other Names: ECLiPS
Behavioral: Multidisciplinary behavioral assessment — By collecting behavioral measures, the investigators wish to understand the functional implications of the presented problems. Children will complete various well-chosen tasks using a tablet, in the presence of a trained clinician. Tablets are used as they are ubiquitous, cost-effective, and have excellent quality audio output. The investigators will apply the concept of differential testing (Dillon & Cameron, 2021; Lagacé et al., 2010) to narrow down the range of deficits that lead to deficient scores. The investigators distinguish four (partly overlapping) categories of behavioral measures: 1) auditory processing, 2) (nonsense) speech sound processing in quiet and in noise, excluding semantics, 3) meaningful speech in quiet and in noise, language processing, and 4) neurocognitive (including attention, memory, processing speed) processing.

SUMMARY:
Many children experience listening and processing difficulties (LiD), especially in background noise, despite normal hearing sensitivity. The prevalence of these problems is estimated at 0.5-1% in the general population. Listening difficulties are associated with developmental disorders (DD) such as specific language disorders, autism spectrum disorder (ASD), ADHD and learning disabilities. Many children with developmental problems are easily distracted by sounds, have difficulty concentrating for long periods, processing language, remembering and summarizing oral information, and can experience academic difficulties (reading, writing). Early identification, differential diagnosis and intervention are important to help children overcome these difficulties and reach their full potential. Some concerns about these listening and processing problems, such as the lack of a gold standard to diagnose LiD and age-appropriate reference data, led to the initiation of this study.

CLINIC aims to develop a new approach to diagnose the causes of listening difficulties in children. This is accomplished through (1) a validated parent questionnaire and (2) a multidisciplinary behavioral assessment tool. Data from these combined measures will lead to evidence-based profiles of children with LiD, which in turn will help streamline their referral pathways and care pathways.

DETAILED DESCRIPTION:
The goal of the CLINIC project is to develop a new approach to diagnose the causes of LiD in 6 to 14-year-old children with normal peripheral hearing. A multicentric, interventional study focuses on the longitudinal evaluation of children with various DDs: SLI, LD, ADHD, and ASS. These children are tested at different sites for three years consecutively with a multidisciplinary behavioral assessment app (CLINIC) that will allow assessing a broad range of skills (auditory abilities, speech processing skills, language abilities, neurocognitive abilities). Profiles of children with LiD will be constructed from the ECLiPS (Evaluation of Children's Listening and Processing Skills; a validated parent report questionnaire) and from the behavioral measures obtained with the CLINIC app, both at a population level and in specialized centers treating children with recognized DD. This will be done in a longitudinal design (3 years) with the same children, to determine age effects and to capture potential changes in the profiles of children with time. Results will be compared with performance of TD children, to determine cut-off criteria for establishing a diagnosis. Comparison of the ECLiPS and the behavioral measures will indicate whether the ECLiPS can be used as a screening measure in the future to help identify children in need of support (and to pinpoint in which domains the support needs to be prioritized).

ELIGIBILITY:
Inclusion Criteria:

* 6 to 14 years old
* experiencing listening difficulties
* normal or near-to-normal hearing (bilateral PTA ≤ 20 dB HL)

Exclusion Criteria:

* acquired conditions (such as brain damage, neuropathy, children with cochlear implants, peripheral hearing loss, or chronic otitis media)
* Down syndrome or another syndrome
* IQ < 70
* hearing loss

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
ECLiPS questionnaire | Year 1, year 2, year 3
  The Evaluation of Children's Listening & Processing Skills (ECLiPS; Barry & Moore, 2021; Barry et al., 2015; Petley et al., 2021) is a caregiver-report outcome measure to profile auditory and cognitive real-world abilities important for successful listening and (auditory) processing.
Behavioral measures | Year 1, year 2, year 3
  Behavioral tasks in different domains (auditory processing, speech processing, language processing, cognition) are administered.